CLINICAL TRIAL: NCT02647294
Title: Nutrition-based Therapy of Liver Disease of Different Origin: Effect of n-3 Polyunsaturated Fatty Acid in Patients With Nonalcoholic Fatty Liver Disease (NAFLD) and Metabolic Syndrome.
Brief Title: Polyunsaturated Fatty Acids in Patients With NAFLD.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Radan Bruha, Clinical associated professor, General University Hospital, Prague
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-28745A
Record Dates: First submitted 2016-01-04; First posted 2016-01-06 (Estimated); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polyunsaturated omega-3 fatty acids (Experimental): Patients will receive n-3 fatty acids (Maxicor) 3,6 g/day.
  Interventions: Dietary Supplement: Maxicor
- Placebo (Placebo Comparator): Patients will receive placebo (soya oil)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Maxicor — Patients with NAFLD will be randomly allocated to receive or n-3 PUFA (3,6 g/day, oral treatment) or placebo (1:1).
  Other Names: n-3 polyunsaturated fatty acids; n-3 PUFA
  Arms: Polyunsaturated omega-3 fatty acids
Other: Placebo — Patients with NAFLD will be randomly allocated to receive or placebo or n-3 PUFA for 12 months (1:1).
  Arms: Placebo

SUMMARY:
Patients with metabolic syndrome and Nonalcoholic fatty liver disease (NAFLD) will be randomly allocated for the treatment with n-3 PUFA (3.6 g/day) or placebo for 12 months. At the beginning and at the end of the study basic clinical and anthropometric data, as well as parameters of liver steatosis and fibrosis will be tested.

DETAILED DESCRIPTION:
Patients with metabolic syndrome and Nonalcoholic fatty liver disease (NAFLD) will be randomly allocated for the treatment with n-3 PUFA (3.6 g/day) or placebo for 12 months. At the beginning and at the end of the study basic clinical and anthropometric data will be recorded and the following parameters will be tested:

panel of biochemistry and liver function tests: triglycerides, cholesterol, HDLcholesterol, LDL-cholesterol, glucose, insulin, serum bilirubin, liver tests, thyroid hormones, bile acids and their metabolites, albumin, total protein.

Bioactive metabolites, Inflammatory markers Non-invasive serum markers of liver fibrosis and steatohepatitis. Hyaluronic acid, NAFLD fibrosis score, cytokeratine-18 fragments. Ultrasonography with non-invasive measurement of fibrosis and steatosis, magnetic resonance spectroscopy for visceral and liver fat determination.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metabolic syndrome and NAFLD

Exclusion Criteria:

* Age below 18 years
* Gravidity
* Incompliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with decreased liver fat content. | 12 months
  Liver fat content in patients will be measured by magnetic resonance before and after the treatment. The number of patients with decreased liver fat content is expected to be higher in the treated group compare to placebo group.

SECONDARY OUTCOMES:
Number of patients with progression of liver fibrosis. | 12 months
  Liver fibrosis will be measured by ultrasound (ARFI) before and after the treatment. The number of patients with no progression of fibrosis is expected to be higher in the treated group compare to placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Radan Bruha, MD, Principal Investigator — General University Hospital, Prague
Locations (1):
- General University Hospital, Prague, Prague 2, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Available upon individual request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Will be available from 6/2023 by the end of 2025.
Access Criteria: Available upon individual request.
URL: https://int4.lf1.cuni.cz/en

REFERENCES:
- [Result] Smid V, Dvorak K, Sedivy P, Kosek V, Lenicek M, Dezortova M, Hajslova J, Hajek M, Vitek L, Bechynska K, Bruha R. Effect of Omega-3 Polyunsaturated Fatty Acids on Lipid Metabolism in Patients With Metabolic Syndrome and NAFLD. Hepatol Commun. 2022 Jun;6(6):1336-1349. doi: 10.1002/hep4.1906. Epub 2022 Feb 11. PMID 35147302